CLINICAL TRIAL: NCT02988752
Title: Comparison Between an Electronic Mobile Device(DEM) and Optical Coherence Tomography (OCT) to Determine Cup-to-disc Ratio (C/D) Through a Non-inferiority Trial With Masked Data Analysis
Brief Title: Comparison Between an Electronic Mobile Device and Optical Coherence Tomography to Determine Cup-to-disc Ratio
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Clinica Oftamologica Zona Sul (Other)
Responsible Party: Principal Investigator, Andrea Gondim Leitao Sarmento, MD, Clinica Oftamologica Zona Sul
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: COZ001
Record Dates: First submitted 2016-06-02; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electronic Mobile Device (Experimental): Use an Electronic Low Cost Mobile Device To Determine C/D Ratio And Compare Results With Gold Standard Optical Coherence Tomography Results. The equipment needs mydriatic conditions and does not touch the patient's eye. The equipment uses a panoptik and a camera to access eye fundus.
  Interventions: Device: Electronic Mobile Device
- Optical Coherence Tomography (Active Comparator): Device considered as gold standard to determine c/d ratio. Needs mydriatic conditions.
  Interventions: Device: Optical Coherence Tomography

INTERVENTIONS:
Device: Electronic Mobile Device — Measure C/D Ratio With An Equipment Attached To A Ophthalmoscope That Will Determine C/D Ratio Without Touching Patient's Eyes. To Perform It We Need Mydriatic Conditions.
  Arms: Electronic Mobile Device
Device: Optical Coherence Tomography — Measure C/D Ratio With OCT, Considered Gold Standard Equipment
  Other Names: OCT
  Arms: Optical Coherence Tomography

SUMMARY:
This study was a non-inferiority trial with masked data analysis. Individuals ranging from 18 to 60 years from both genders that met the pre-defined criteria were included. This study was carried out in Recife at Clinica Oftalmologica Zona Sul and at Centro de Informatica-UFPE. Using both equipment, 5 vertical cup-to-disc ratio (VCDR) evaluations were performed for each eye of the individuals, under midriatic conditions. Evaluations were done by examiners who did not know previously results obtained from other equipment. Data was collected by the main researcher of this research. This study was approved by the ethics committee before it started and all research members signed the TCLE agreement. The statistical test employed in this study was Pearson Correlation test.

DETAILED DESCRIPTION:
Glaucoma is the second major cause of blindness in the world, lagging only behind cataract. However, unlike cataract, blindness caused by glaucoma is irreversible. Early diagnosis of the disease and progression monitoring is thus essential for proper treatment in order to avoid irreversible blindness. The most common screening exam for glaucoma diagnosis and monitoring is the eye fundus evaluation where Cup-to-Disc ratio (CDR) among other parameters are assessed. This kind of evaluation is performed by ophthalmologists based on their visual perception, requiring not only specific training but also some significant amount of time of eye examination.Objective measurement of CDR involves high cost equipment which in turn requires some specific training in order to use them. Currently, the Optical Coherence Tomography is used as the gold standard for CDR measurement. An OCT exam uses a high cost and complex equipment that most of the time is not affordable for low-income people. This study proposes a portable electronic device that captures eye fundus images, analyzes these images, performs CDR calculation and allows storing these images for further analysis. This low cost and portable device was developed to be used in several health services (public or private) and has low energy consumption, easing its mobility. Moreover, using this device is easy, not requiring any significant learning effort from ophthalmologists. In developing countries where screening programs for early diagnosis of glaucomatous neuropathy are adopted, an ever-growing number of researchers are putting a significant amount of effort to develop cost-benefit solutions that can reach low-income people and remote areas.

Objective: This study compared CDR measurements from the portable electronic device (PED) developed by Centro de Informatica da Universidade Federal de Pernambuco to CDR measurements provided by OCT.

Methods:This study was a non-inferiority trial with masked data analysis. Individuals ranging from 18 to 60 years from both genders that met the pre-defined criteria were included. This study was carried out in Recife at Clinica Oftalmologica Zona Sul and at Centro de Informatica-UFPE. Using both equipment, 5 vertical cup-to-disc ratio (VCDR) evaluations were performed for each eye of the individuals, under midriatic conditions. Evaluations were done by examiners who did not know previously results obtained from other equipment. Data was collected by the main researcher of this research. This study was approved by the ethics committee before it started and all research members signed the TCLE agreement. The statistical test employed in this study was Pearson Correlation test.

ELIGIBILITY:
Inclusion Criteria:

* Anyone from 18 to 60 Years old without any of the Specified Exclusion Criteria.

Exclusion Criteria:

* Cancer
* Cataract
* Eyes transparency loss
* Best Av < 0.4
* Eye surgery in the last 12 Months
* Use of drugs that leads to any kind of Neuropathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Objective C/D Ratio measure | One Year
  To measure vertical cup to disc ratio in an objective way

CONTACTS AND LOCATIONS:
Overall Officials: ANDREA SARMENTO, Principal Investigator — COZ
Locations (1):
- Clinica Oftalmologica Zona Sul, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No